CLINICAL TRIAL: NCT02539446
Title: The Effects of Suprapostural Attention Focus and Postural Difficulty on H-reflex and Brain Activity: Aging and Parkinson's Disease
Brief Title: Suprapostural Attention Focus and Postural Difficulty on H-reflex and Brain Activity: Aging and Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 201312077RINC
Record Dates: First submitted 2014-10-21; First posted 2015-09-03 (Estimated); Last update posted 2019-12-16 (Actual); Status verified 2016-10

CONDITIONS: Parkinson
Keywords: Aging; External focus; Internal focus; Attention; Posture balance; Parkinson's disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- stable condition & attentional focus (Other): for measure the relationships between task difficulty and attentional focus on supraposture
  Interventions: Behavioral: stable condition; Behavioral: attentional focus
- unstable condition & attentional focus (Other): for measure the relationships between task difficulty and attentional focus on supraposture
  Interventions: Behavioral: unstable condition; Behavioral: attentional focus

INTERVENTIONS:
Behavioral: stable condition
  Arms: stable condition & attentional focus
Behavioral: unstable condition
  Arms: unstable condition & attentional focus
Behavioral: attentional focus
  Other Names: internal focus; external focus

SUMMARY:
Inherent with intricate allocation of brain resource and attention shift, postural-suprapostural task is defined as postural control takes place while the other concurrent task is being performed. Recent studies have indicated that attentional focusing alters attention allocation in the brain as well as motor performance of a postural-suprapostural task. Also, most studies have demonstrated benefits of inducing an external focus relative to internal focus for motor performance. However, postural difficulty might be a critical factor for choosing an appropriate focusing strategy, and the strategy used in a particular difficulty level do not always generalize to other difficulty levels. Besides, despite a lot of studies have been done, current findings are confined to behavioral observations in young healthy adults for lacking direct neural evidence. With the uses of H-reflex, event-related potential and behavioral measures, the purpose of the 3-year research project is to investigate the differences in performance quality and intrinsic neural mechanisms of a postural-suprapostural task for older adults and patients with Parkinson's disease, by adopting external and internal strategies for suprapostural task under different posture difficulties. In the first year, the investigators will characterize suprapostural focusing effect on reciprocity of a postural-suprapostural task, with a special focus on modulation of motoneuron excitability in sitting and standing posture for healthy young and older adults using H-reflex technique. In the second year, the adaptive selection of suprapostural focusing strategy will be investigated for patients with Parkinson's disease by varying the standing surface (stable/unstable surface). In the third year, the investigators will investigate suprapostural focusing effect on brain resource allocation for patients with Parkinson's disease, in light of event-related potential and movement-related potential. The present project is expected to have significant contributions not only to gain a better insight to neural correlates of concurrent postural and motor suprapostural tasks with internal/external focusing strategy under different posture difficulty, but to optimize treatment strategy for older adults and patients with Parkinson's disease with balance or multi-tasking disturbances.

ELIGIBILITY:
Inclusion criteria

* Independent standing balance on air pillow at least 20 sec
* No neurologic or orthopedic disorder

Exclusion criteria

* Had relative experience before
* Pregnant women

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-10; Primary Completion 2014-10 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
H-reflex analysis | 1 week
  The value of soleus H/Mmax ratio is measured as the motoneuron excitability

SECONDARY OUTCOMES:
EMG analysis | 1 week
  The root mean square value of right biceps EMG is measured as the muscle activity
postural sway analysis | 1 week
  The root mean square value of center of pressure in anterior-posterior and medial-lateral directions are used as the postural performance

CONTACTS AND LOCATIONS:
Overall Officials: Cheng-Ya Huang, Principal Investigator — National Taiwan University
Locations (2):
- Taiwan (2):
  - National Taiwan University Hospital, Taipei
  - School and Graduate Institute of Physical Therapy, College of Medicine, National Taiwan University, Taipei

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yu SH, Wu RM, Huang CY. Attentional Resource Associated With Visual Feedback on a Postural Dual Task in Parkinson's Disease. Neurorehabil Neural Repair. 2020 Oct;34(10):891-903. doi: 10.1177/1545968320948071. Epub 2020 Aug 24. PMID 32830603
- [Derived] Huang CY, Chen YA, Hwang IS, Wu RM. Improving Dual-Task Control With a Posture-Second Strategy in Early-Stage Parkinson Disease. Arch Phys Med Rehabil. 2018 Aug;99(8):1540-1546.e2. doi: 10.1016/j.apmr.2018.02.013. Epub 2018 Mar 31. PMID 29608901